CLINICAL TRIAL: NCT06185062
Title: Pelvic and Thoracic Cancer Treated With Online Adapted Radiotherapy: A Prospective Registry-based Phase-II Trial
Brief Title: Pelvic Cancer Registry for Online Adapted Radiotherapy
Acronym: PRoART
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Rami El Shafie, Clinical Study Management on behalf of the Principal Investigator, University Medical Center Goettingen
Other Study IDs: 2023-02727
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Pelvic Tumor; Thoracic Tumor
Keywords: online Adaptive Radiotherapy
MeSH Terms: conditions — Pelvic Neoplasms; Thoracic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- oART: Patients with pelvic or thoracic tumors with an indication for radiotherapy treated with oART (online Adaptied Radiotherapy).
- IGRT: Patients with pelvic or thoracic tumors with an indication for radiotherapy treated with conventional IGRT (Image Guided Radiotherapy).

SUMMARY:
This prospective registry-based trial will include patients with pelvic or thoracic tumors with an indication for radiotherapy treated with oART or IGRT. For the primary endpoint and the secondary clinical endpoints, the trial will compare oART versus IGRT, for technical endpoints the trial will compare the real oART scenario with two virtual (hypothetical) control scenarios.

Primary endpoint:

* 10% reduction in the rate of acute radiotherapy related toxicity (≥ CTCAE II°, v5.0) using oART

Secondary endpoints:

* Clinical endpoints: Tumor control, late toxicities compared to conventional irradiated patients, quality of life and patient-reported outcomes
* Technical endpoints: Target volume, target coverage, dose to organs at risk, anatomical variability score

DETAILED DESCRIPTION:
Background: Conventional Radiotherapy (Image Guided Radiotherapy, IGRT) requires a CT-based treatment planning process a priori. During this process, a treatment plan is calculated, which then is applied to the patient with a linear accelerator on a daily basis, possibly using image guidance to account for variability in patient position. However, daily changes of the anatomy of targets and organs at risk (OARs) can only be addressed by applying additional safety margins, resulting in larger irradiated volumes and possibly higher toxicity.

A promising and innovative technique for margin and in consequence toxicity reduction is online Adaptive Radiotherapy (oART) using daily imaging to create a "plan of the day" aligned to the actual anatomy by means of artificial intelligence (AI) and with the patient on the treatment couch. This approach is especially promising in the pelvic region due to the high anatomic variability, e.g. caused by peristalsis or volume changes of bladder and rectum. Furthermore, the application of oART in the field of thoracic tumors is being evaluated. oART is an already established form of treatment which is used regulary everyday in clinical practice and is not a study-related intervention. A direct comparison of both techniques IGRT vs. oART is missing.

Methods: This prospective and retrospective registry-based trial will include patients with pelvic or thoracic tumors with an indication for radiotherapy treated with oART or IGRT. For the primary endpoint and the secondary clinical endpoints, the trial will compare oART versus IGRT, for technical endpoints the trial will compare the real oART scenario with two virtual (hypothetical) control scenarios as follows:

* oART - Applied treatment: AI-based daily treatment plan creation, adapted to daily anatomy
* Virt 1 - Hypothetical dose distribution of initial treatment plan, based on the initial planning CT
* Virt 2 - Hypothetical dose distribution of initial treatment plan, applied to the anatomy of the day as depicted by cone-beam CT at the treatment machine

ELIGIBILITY:
INCLUSION CRITERIA

* Patients with pelvic or thoracic tumors with an indication for radiotherapy
* Patient information and declaration of consent
* Patients age ≥ 18 years

EXCLUSION CRITERIA

* Prior radiotherapy in affected site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients with pelvic or thoracic tumors with an indication for radiotherapy treated with oART or IGRT.
Sampling Method: Non-Probability Sample
Enrollment: 846 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Rate of acute radiotherapy related toxicity | until 12 weeks post RT
  10% reduction in the rate of acute radiotherapy related toxicity (≥ CTCAE II°, v5.0) using oART

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, Departement of Radiation Oncology, Göttingen, Germany